CLINICAL TRIAL: NCT05488431
Title: Cholesterol and Inflammation Lowering Via Bempedoic Acid, an ACL-inhibiting Regimen in HIV Trial (CLEAR HIV Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Priscilla Hsue, MD (Other)
Collaborators: University of California, Los Angeles (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Priscilla Hsue, MD, Dr. Priscilla Hsue, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2022-07-25; First posted 2022-08-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemias; Cardiovascular Diseases; HIV Infections; Atherosclerosis
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; HIV Infections; Atherosclerosis | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bempedoic acid (BA) (Experimental): Patients randomized into the BA arm will receive 180 mg BA administered orally once daily without food for 52 weeks.
  Interventions: Drug: Bempedoic acid
- Placebo (Placebo Comparator): Patients randomized into the placebo arm will receive 180 mg placebo administered orally once daily without food for 52 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bempedoic acid — Bempedoic Acid is an oral first-in-class small molecular adenosine triphosphate (ATP)-citrate lyase (ACL) inhibitor which lowers LDL-C by inhibition of cholesterol synthesis in the liver. ACL is an enzyme upstream of 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase in the cholesterol biosynthesis pathway. Inhibition of ACL by bempedoyl-CoA results in decreased cholesterol synthesis in the liver and lowers LDL-C in blood via upregulation of LDL receptors and concomitant suppression of hepatic fatty acid biosynthesis. BA has been studied in >4300 individuals and is currently being studied in >14,000 individuals in CLEAR Outcomes (NCT02993406).
  Other Names: BA
  Arms: Bempedoic acid (BA)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized placebo-controlled study in treated and suppressed HIV-infected individuals aged ≥40 years with either known CVD or 1 CVD risk factor to study the effect of Bempedoic acid (BA) on safety, arterial inflammation as assessed by FDG-PET/CT, lipids, inflammation, immune activation, cardiometabolic indices, and non-calcified plaque (NCP) in the coronary arteries (assessed by coronary CT angiography, CCTA). This trial will be enrolled at UCSF and UCLA. Collaborators at Massachusetts General Hospital (MGH) will serve as the core facility for imaging.

DETAILED DESCRIPTION:
Persons living with HIV infection (PLWH) have a 2-fold higher risk of myocardial infarction and are twice as likely to develop cardiovascular disease accounting for a significant global burden of disease. While the mechanism underlying this excess risk remains poorly understood, studies demonstrate that atherosclerosis in the setting of HIV is distinct and characterized by heightened arterial inflammation as assessed by FDG-PET/CT. HIV and antiretroviral medication can worsen cardiometabolic parameters. Thus a therapeutic strategy that can lower lipids, inflammation, and improve glycemic parameters may be even more advantageous in HIV. Bempedoic acid (BA, an inhibitor of ATP citrate lyase), is safely tolerated, significantly lowers LDL-C and inflammatory markers (on top of statin therapy), and is FDA approved for individuals with heterozygous familial hypercholesterolemia or with established ASCVD who require additional LDL-C lowering. Additionally, BA has a protective effect on glycemic parameters and may reduce adiposity. Given the key role of lipids and inflammation in atherosclerosis in HIV, the purpose of this proof-of-concept mechanistic trial is to evaluate the impact of BA on the biology of HIV-associated atherosclerosis. This is a randomized placebo controlled study of effectively treated PLWH aged 40 years and older with either known CVD or 1 CVD risk factor to study the effect of BA on arterial inflammation (assessed by FDG-PET/CT), lipid levels, biomarkers of inflammatory/immune activation, cardiometabolic indices, and non-calcified plaque in the coronary arteries (assessed by CCTA). This multicenter trial will include PLWH enrolled at UCSF and UCLA. Long term collaborators at MGH will serve as the core facility for the imaging end-points. There are three specific aims for the: Cholesterol and inflammation Lowering via BEmpedoic Acid, an ACL-inhibiting Regimen in HIV Trial (CLEAR HIV Trial): Aim 1: To determine whether BA can safely reduce arterial inflammation including carotid plaque as assessed by FDG-PET/CT; Aim 2: To determine whether BA improves cardiometabolic measures (lipid, inflammatory, glycemic and adipose parameters) among PLWH. Exploratory objectives will be to assess BA's effect (vs. placebo) on glycemic as well as adipose tissue measures (HbA1c, HOMA IR, and adipose tissue volumes); Aim 3: To evaluate the impact of BA on non-calcified coronary plaque volume as measured by coronary CT angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* On continuous antiretroviral therapy and virologically suppressed HIV infection for ≥12 weeks prior to study entry
* CD4 T-cell count ≥ 200 cells/mm3
* Male or female between the ages ≥ 40 years of age
* LDL-C ≥ 50 mg/dL
* Documented cardiovascular disease as defined by: 1. Prior myocardial infarction, 2. Prior cerebrovascular disease, 3. Prior peripheral arterial disease, 4. History of percutaneous coronary intervention, 5. History of coronary artery bypass graft OR 6. Angiographic evidence of >50% stenosis in at least one coronary artery] OR 1 CVD risk factor (T2DM, current smoking, hypertension, dyslipidemia, hsCRP≥2mg/L, family history)
* TBR of >1.6 of the MDS of the carotid/aorta at baseline. This baseline arterial TBR cutoff excludes the rare individual that lacks appreciable arterial inflammation. It is notable that while 5-10% of uninfected individuals will have lower TBRs, it is rare that an HIV infected individual will fall below this range.
* Female subjects must either be of non-childbearing potential (defined as post-menopausal or amenorrhea > 12 months) or agree to use two forms of contraception (one hormonal and one barrier) throughout the study and for at least one month following study completion and have a negative pregnancy test at screening and prior to the first dose of drug.
* Males must use at least one method of contraception throughout the study.

Exclusion Criteria:

* Pregnant/nursing women (as there is no data on bempedoic acid in this setting)
* Diabetes requiring insulin (as insulin treatment alters the uptake of 18FDG)
* Uncontrolled HTN as defined by baseline blood pressure reading of ≥160 mmHg systolic OR ≥100 mmHg diastolic (exclusion criteria in other studies with BA)
* AST/ALT or alkaline phosphatase >2x ULN
* Triglycerides >500 mg/dL at screening
* Cancer within the last 5 years with exception of squamous cell carcinoma and basal cell carcinoma
* Individuals on simvastatin >20mg or pravastatin >40mg. All other dosages and statins will be permitted with close monitoring for myopathies including assessment of CK levels
* Nephrotic syndrome or eGFR <30 mL/min/1.73m2
* Cytopenias which include 1) WBC <3.5 x103/uL 2) Platelet <120 x103/uL 3) ANC <1.5 x103/uL, and absolute lymphocytes <0.8 x 103/uL
* Anemia as fined by Hgb <10 g/dL
* Acute systemic infection within 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
FDG PET/CT Endpoint | Baseline and Week 52
  Change in Target-to-background ratio from baseline to follow-up study at 52 weeks. The main arterial endpoint is the most diseased segment of the index vessel. These findings will be correlated to measurements in the secondary endpoint.

SECONDARY OUTCOMES:
Total Cholesterol Endpoint | Baseline, Week 24 and Week 52
  Change in total cholesterol will be assessed from baseline to week 24 and week 52.
HDL Endpoint | Baseline, Week 24 and Week 52
  Change in HDL will be assessed from baseline to week 24 and week 52.
LDL Endpoint | Baseline, Week 24 and Week 52
  Change in LDL will be assessed from baseline to week 24 and week 52.
Triglycerides Endpoint | Baseline, Week 24 and Week 52
  Change in triglycerides will be assessed from baseline to week 24 and week 52.
Apolipoprotein B Endpoint | Baseline, Week 24 and Week 52
  Change in apolipoprotein B will be assessed from baseline to week 24 and week 52.
Hb A1c Endpoint | Baseline, Week 24 and Week 52
  Change in HbA1c from baseline to week 24 and week 52.
Fasting glucose Endpoint | Baseline, Week 24 and Week 52
  Change in fasting glucose measurements from baseline to week 24 and week 52.
Insulin Endpoint | Baseline, Week 24 and Week 52
  Change in insulin measurements from baseline to week 24 and week 52.
homeostatic Model Assessment for Insulin Resistance (HOMA-IR) Endpoints | Baseline, Week 24 and Week 52
  The change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), a calculation based on insulin and glucose, will also be assessed from baseline to week 24 and 52.
  The equation simplifies to [HOMA-IR = fasting insulin *fasting glucose /22.5] where fasting plasma insulin is measured in (µIU/mL) and fasting plasma glucose is measured in (mmol/L). Values below 1.0 are generally considered optimal.
Adipose Volume Endpoint | Baseline and Week 52
  Change in adipose tissue volumes will be assessed by FDG PET/CT (as measured in primary outcome) from baseline to week 52.
hsCRP Endpoint | Baseline, Week 24 and Week 52
  Change in hsCRP from baseline to follow-up at weeks 24 and 52.
IL-1B Endpoint | Baseline, Week 24 and Week 52
  Change in IL-1B from baseline to follow-up at weeks 24 and 52.
IL-18 Endpoint | Baseline, Week 24 and Week 52
  Change in IL-18 from baseline to follow-up at weeks 24 and 52.
SAA Endpoint | Baseline, Week 24 and Week 52
  Change in SAA from baseline to follow-up at weeks 24 and 52.
Lp-PLA2 Endpoint | Baseline, Week 24 and Week 52
  Change in Lp-PLA2 from baseline to follow-up at weeks 24 and 52.
sCD163 Endpoint | Baseline, Week 24 and Week 52
  Change in sCD163 from baseline to follow-up at weeks 24 and 52.
IL-6 Endpoint | Baseline, Week 24 and Week 52
  Change in IL-6 from baseline to follow-up at weeks 24 and 52.
D-Dimer Endpoint | Baseline, Week 24 and Week 52
  Change in D-Dimer from baseline to follow-up at weeks 24 and 52.
Fibrinogen Endpoint | Baseline, Week 24 and Week 52
  Change in fibrinogen from baseline to follow-up at weeks 24 and 52.
T-cell Endpoint | Baseline, Week 24 and Week 52
  Change in T-cell marker from baseline to follow up at weeks 24 and 52.
B-cell Endpoint | Baseline, Week 24 and Week 52
  Change in B-cell marker from baseline to follow up at weeks 24 and 52.
Monocyte activation Endpoint | Baseline, Week 24 and Week 52
  Change in monocyte activation marker from baseline to follow up at weeks 24 and 52.

OTHER OUTCOMES:
Coronary CTA Non-calcified Plaque Endpoint | Baseline and Week 52
  Change in non-calcified plaque as measured by Coronary CTA from baseline to follow-up study at 52 weeks
Coronary CTA High-risk Plaque Endpoint | Baseline and Week 52
  Change in high-risk plaque as measured by Coronary CTA from baseline to follow-up study at 52 weeks.
Coronary CTA Coronary Plaque Incidence Endpoint | Baseline and Week 52
  Incidence of new coronary lesions as measured by Coronary CTA from baseline to follow-up study at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - UCLA Center for Clinical AIDS Research and Education (CARE), Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No